CLINICAL TRIAL: NCT01093014
Title: Novel Intervention to Influence Muscle Plasticity in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7097-R
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injuries
Keywords: Quadriceps Muscle; RNA, Messenger; Hypertrophy; Electric Stimulation Therapy
MeSH Terms: conditions — Spinal Cord Injuries; Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: High-force muscle stimulation (Experimental): High-force muscle stimulation
  Interventions: Behavioral: High-force muscle stimulation
- Arm 2: Low-force muscle stimulation (Experimental): Low-force muscle stimulation
  Interventions: Behavioral: Low-force muscle stimulation
- Arm 3: Sequential low-force and high-force muscle stimulation (Experimental): Sequential low-force and high-force muscle stimulation
  Interventions: Behavioral: Sequential low-force and high-force muscle stimulation

INTERVENTIONS:
Behavioral: Low-force muscle stimulation — Electrical stimulation of paralyzed muscle in seated or standing to evoke non-summated, low-force contractions, using either a lab-based system or a portable system for up to 1 year.
  Arms: Arm 2: Low-force muscle stimulation
Behavioral: High-force muscle stimulation — Electrical stimulation of paralyzed muscle in seated or standing to evoke summated, high-force contractions, using either a lab-based system or a portable system for up to 1 year.
  Arms: Arm 1: High-force muscle stimulation
Behavioral: Sequential low-force and high-force muscle stimulation — Electrical stimulation of paralyzed muscle in seated or standing to evoke non-summated, low-force contractions, followed by: 1) a 1-month washout period, then; 2) electrical stimulation to evoke summated, high-force contractions.
  Arms: Arm 3: Sequential low-force and high-force muscle stimulation

SUMMARY:
The loss of muscle contraction (paralysis) removes an important stimulus for maintenance of overall health for individuals with complete spinal cord injury (SCI). Increased protein catabolism (atrophy) limits important stresses to the skeletal system. Bone loss doubles the risk of fracture and contributes to increased mortality in Veterans with SCI. Metabolic syndrome and diabetes lead to heart disease in Veterans with SCI at higher rates than the general population. Exercise methods to sustain muscle tissue, bone density, and metabolic stability after SCI are lacking scientific justification. If left unchecked, the secondary complications of SCI can be health limiting or even life threatening to Veterans with paralysis. The importance of maintaining the health of the musculoskeletal system after SCI has never been greater as a cure for paralysis may become a reality. Contemporary rehabilitation interventions lack the ability to functionally load muscle tissue, quantify the dose of load, stress the cardiovascular system, monitor the overall stresses during daily exercise training, or offer portability to improve compliance with the exercise. The long-term goal of this project is to establish the optimal dose of muscle and bone stress during functional exercise in order to improve the health of Veterans with complete paralysis. The practical outcome of this research is to offer a form of activity that is feasible, portable, and grounded in sound scientific principles. The scientific goal is to understand whether the dose of force generated in paralyzed muscle via evoked contractions is critical to muscle atrophy/hypertrophy molecular pathways, physiologic performance, and insulin sensitivity. The investigators will administer various doses of muscle force by manipulating the frequency of electrical stimulation while keeping stimulation current (i.e. muscle fiber recruitment) constant. Interestingly, no previous study has examined the dose of muscle force necessary to trigger adaptations in protein synthesis/degradation pathways. The investigators wish to discover the most effective method to maintain the molecular and physiologic properties of paralyzed muscle. The investigators believe such a method will be in urgent demand as a co-intervention with pharmaceutical strategies in post-SCI rehabilitation.

DETAILED DESCRIPTION:
Central Hypothesis: The investigators hypothesize that high muscle force induced via a novel, portable, active standing intervention will increase muscle force properties, alter gene expression for atrophy and fiber type pathways, and improve systemic insulin sensitivity in Veterans with complete paralysis.

Aim 1: To determine the training effects of 3 tiers of quadriceps muscle force on muscle physiological properties in Veterans with chronic paralysis from SCI.

Aim 2: To determine the training effects of 3 tiers of quadriceps muscle forces on muscle mRNA for genes associated with atrophy and muscle fiber type in Veterans with complete paralysis.

Aim 3: To determine the training effects of 2 tiers of compressive load induced by quadriceps muscle forces on insulin sensitivity and markers of inflammation in Veterans with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for all subjects will be upper motor neuron lesions between the 10th thoracic and the 7th cervical spinal levels. The completeness of the injury will be verified by somatosensory evoked potentials.

Exclusion Criteria:

* Subjects will be excluded if they have pressure ulcers
* chronic infection
* lower extremity muscle contractures
* deep vein thrombosis
* recent limb fractures
* muscle metabolic disorders
* any comorbid disease known to affect bone metabolism (such as parathyroid dysfunction)
* or if they are pregnant or plan to become pregnant.
* Subjects with distal femur trabecular bone mineral density less than 50 mg/cm3 will be excluded from participation in quadriceps electrical stimulation training

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Shields, PhD PT, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams CM, Suneja M, Dudley-Javoroski S, Shields RK. Altered mRNA expression after long-term soleus electrical stimulation training in humans with paralysis. Muscle Nerve. 2011 Jan;43(1):65-75. doi: 10.1002/mus.21831. PMID 21171097
- [Background] Kunkel SD, Suneja M, Ebert SM, Bongers KS, Fox DK, Malmberg SE, Alipour F, Shields RK, Adams CM. mRNA expression signatures of human skeletal muscle atrophy identify a natural compound that increases muscle mass. Cell Metab. 2011 Jun 8;13(6):627-38. doi: 10.1016/j.cmet.2011.03.020. PMID 21641545
- [Background] McHenry CL, Shields RK. A biomechanical analysis of exercise in standing, supine, and seated positions: Implications for individuals with spinal cord injury. J Spinal Cord Med. 2012 May;35(3):140-7. doi: 10.1179/2045772312Y.0000000011. PMID 22507023
- [Background] Dudley-Javoroski S, Shields RK. Regional cortical and trabecular bone loss after spinal cord injury. J Rehabil Res Dev. 2012;49(9):1365-76. doi: 10.1682/jrrd.2011.12.0245. PMID 23408218
- [Result] Dudley-Javoroski S, Saha PK, Liang G, Li C, Gao Z, Shields RK. High dose compressive loads attenuate bone mineral loss in humans with spinal cord injury. Osteoporos Int. 2012 Sep;23(9):2335-46. doi: 10.1007/s00198-011-1879-4. Epub 2011 Dec 21. PMID 22187008
- [Result] Petrie MA, Suneja M, Faidley E, Shields RK. Low force contractions induce fatigue consistent with muscle mRNA expression in people with spinal cord injury. Physiol Rep. 2014 Feb 25;2(2):e00248. doi: 10.1002/phy2.248. eCollection 2014 Feb 1. PMID 24744911
- [Result] Petrie MA, Suneja M, Faidley E, Shields RK. A minimal dose of electrically induced muscle activity regulates distinct gene signaling pathways in humans with spinal cord injury. PLoS One. 2014 Dec 22;9(12):e115791. doi: 10.1371/journal.pone.0115791. eCollection 2014. PMID 25531450
- [Result] Petrie M, Suneja M, Shields RK. Low-frequency stimulation regulates metabolic gene expression in paralyzed muscle. J Appl Physiol (1985). 2015 Mar 15;118(6):723-31. doi: 10.1152/japplphysiol.00628.2014. Epub 2015 Jan 29. PMID 25635001

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: High-force Muscle Stimulation | Arm 2: Low-force Muscle Stimulation | Arm 3: Sequential Low-force and High-force Muscle Stimulation
Started | 12 | 9 | 12
Completed | 12 | 9 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: High-force Muscle Stimulation | Arm 2: Low-force Muscle Stimulation | Arm 3: Sequential Low-force and High-force Muscle Stimulation | Total
Number analyzed (Participants) | 12 | 9 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.33 (7.45) | 36.0 (32.3) | 32.3 (9.1) | 32.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 8
  Male | 9 | 6 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: HF Muscle Force
Description: Muscle force evoked during high-force muscle stimulation
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: Newtons (N)
Groups:
- Arm 1: High-force Muscle Stimulation: High-force muscle stimulation: Electrical stimulation of paralyzed muscle to evoke summated, high-force contractions, using either a lab-based system or a portable system for up to 1 year.
- Arm 2: Low-force Muscle Stimulation: Low-force muscle stimulation: Electrical stimulation of paralyzed muscle to evoke non-summated, low-force contractions, using either a lab-based system or a portable system for up to 1 year.
- Arm 3: Sequential Low-force and High-force Muscle Stimulation: Sequential low-force and high-force muscle stimulation: Electrical stimulation of paralyzed muscle to evoke non-summated, low-force contractions, followed by: 1) a 1-month washout period, then; 2) electrical stimulation to evoke summated, high-force contractions.
Arm/Group | Arm 1: High-force Muscle Stimulation | Arm 2: Low-force Muscle Stimulation | Arm 3: Sequential Low-force and High-force Muscle Stimulation
Number analyzed (Participants) | 12 | 0 | 12
Newtons (N) | 23.9 (5.9) |  | 30.9 (5.5)

2. Primary Outcome: LF Muscle Force
Description: Muscle force evoked during low-force muscle stimulation
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: N (newtons)
Arm/Group | Arm 1: High-force Muscle Stimulation | Arm 2: Low-force Muscle Stimulation | Arm 3: Sequential Low-force and High-force Muscle Stimulation
Number analyzed (Participants) | 0 | 9 | 12
N (newtons) |  | 26.72 (19.03) | 27.58 (4.41)

3. Primary Outcome: Skeletal Muscle Gene Regulation: MSTN
Description: Messenger ribonucleic acid (mRNA) expression fold-change for myostatin (MSTN). Fold change: post-intervention expression / pre-intervention expression. Values greater than 1.0 indicate up-regulation. Values less than 1.0 indicate down-regulation.
Time Frame: up to 1 year
Population: Only a subset of Arm 1 and Arm 3 participants underwent biopsy: we achieved statistical power with these subsets and further biopsies were not warranted.
Measure: Mean (Standard Deviation); unit: fold-change
Arm/Group | Arm 1: High-force Muscle Stimulation | Arm 2: Low-force Muscle Stimulation | Arm 3: Sequential Low-force and High-force Muscle Stimulation
Number analyzed (Participants) | 3 | 0 | 6
fold-change | .56 (.06) |  | .67 (.40)

4. Primary Outcome: Skeletal Muscle Gene Expression: PPARGC1A
Description: Messenger ribonucleic acid (mRNA) expression fold-change for peroxisome proliferator-activated receptor gamma, coactivator 1 alpha (PPARGC1A). Fold change: post-intervention expression / pre-intervention expression. Values greater than 1.0 indicate up-regulation. Values less than 1.0 indicate down-regulation.
Time Frame: up to 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: fold-change
Arm/Group | Arm 1: High-force Muscle Stimulation | Arm 2: Low-force Muscle Stimulation | Arm 3: Sequential Low-force and High-force Muscle Stimulation
Number analyzed (Participants) | 3 | 0 | 6
fold-change | 5.46 (.64) |  | 4.97 (3.5)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Arm 1: High-force Muscle Stimulation | Arm 2: Low-force Muscle Stimulation | Arm 3: Sequential Low-force and High-force Muscle Stimulation
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes